CLINICAL TRIAL: NCT02302924
Title: Evaluation of Psychometric Testing Properties of Severity Symptom Grading Scale of Influenza Infection: Flu-PRO Stage III
Acronym: FluPRO3
Status: Completed | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Evidera (Industry); Leidos Biomedical Research, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IDCRP-081
Record Dates: First submitted 2014-11-24; First posted 2014-11-27 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Influenza; Influenza-like Illness
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — After obtaining informed consent, an oral/nasal swab or wash to confirm or rule out an influenza etiology will be collected at baseline if the participant does not already have documented laboratory confirmation of influenza.
Oversight: Data Monitoring Committee: No

SUMMARY:
There is no standardized method for evaluating the symptoms of influenza. A standardized instrument for measuring influenza symptoms, with appropriate scientifically derived content and construct validity would have value for public health in terms of use as a validated outcome measure in interventions to treat or prevent influenza. The instrument also could serve as part of an overall measure of severity of illness in influenza. Previous efforts in participant reported outcomes (PRO) for influenza (i.e. Flu-PRO Stage I and Stage II) focused on the elicitation and evaluation of items for inclusion in the instrument. The overarching objective of this protocol - Flu-PRO Stage III - is to conduct instrument validation to evaluate item properties and, if need be, reduce the number of items, and quantitatively validate the performance of the final measure.

DETAILED DESCRIPTION:
The overarching purpose of this study is to develop a single, standardized measurement scale of participant influenza symptoms for use in clinical studies involving adult and pediatric participants. The development of an instrument for participant reported outcomes of influenza was composed of three stages, as described below:

Stage I. Elicitation interviews in a group of volunteers with laboratory-confirmed influenza to inform the development of the instrument, including its content and structure (item phrasing, length, response options, recall).

Stage II. Evaluative interviews with a second set of volunteers with laboratory-confirmed influenza to assess comprehension and interpretability of the instrument and draft item pool from the respondent's perspective.

Stage III. Item reduction and instrument validation in a third set of volunteers to evaluate item properties and quantitatively validate the performance of the final measure.

This protocol will describe the rationale, design, data collection procedures, and analysis methods for Stage III - Item Reduction and Instrument Validation.

ELIGIBILITY:
Inclusion Criteria:

* DEERS eligible
* Adults ≥18 years
* Influenza or influenza-like symptoms as defined by one or more of the following:

  * Positive influenza test by PCR, culture, and/or rapid antigen testing
  * Fever with temperature ≥100.4° F [38° C] AND Respiratory Symptoms* OR
  * Subjective fever AND Respiratory Symptoms* [*Respiratory Symptoms: cough, or sputum production, or shortness of breath, or chest pain, and/or sore throat]
* Speak and read English
* Access to the internet through computer, laptop, tablet, or smartphone

Exclusion Criteria:

* Individuals who do not have access to the internet by computer, laptop, tablet, or smartphone
* Individuals with cognitive and/or physical disabilities who are unable to use a touch screen or computer mouse to enter information into an internet-based survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The targeted sample population will be recruited from the United States. Participants at the IDCRP sites will be both male and female military health care beneficiaries age 18 years and older presenting with the diagnosis of influenza or with influenza-like symptoms suggestive of infection.
Sampling Method: Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The purpose of Flu-PRO Stage III is to conduct a quantitative validation of the FLU-PRO instrument to assess its performance as a standardized method to evaluate symptoms of influenza in natural history studies and clinical trials. | 1 year
  The study will utilize a prospective design to enroll participants with laboratory-confirmed influenza and to capture information regarding the severity of symptoms. This data will be used to validate the Flu-PRO instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Fairchok, MD, Principal Investigator — Madigan Army Medical Center
Locations (5):
- United States (5):
  - Naval Medical Center San Diego, San Diego, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Brooke Army Medical Center, San Antonio, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - Madigan Army Medical Center, Tacoma, Washington